CLINICAL TRIAL: NCT04090307
Title: Targeted Lifestyle Change (TLC) Group Prenatal Care for Obese Women at High Risk for Gestational Diabetes: a Randomized Controlled Trial
Brief Title: Targeted Lifestyle Change Group Prenatal Care
Acronym: TLC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23-2333
Record Dates: First submitted 2019-08-09; First posted 2019-09-16 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy; Gestational Diabetes
Keywords: Group Prenatal Care; Diabetes
MeSH Terms: conditions — Diabetes, Gestational; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TLC Group Prenatal Care (Experimental): TLC will start in the late first trimester or early second trimester and run for ~6-10 sessions. Groups of 2-10 consented women, with two or more GDM risk factors, will meet under the supervision of an obstetric provider (nurse practitioner or MD) and co-facilitator (health educator, nutritionist, or nurse) for two-hour sessions. A major focus of TLC will be education, and much of each visit will be spent on pregnancy, exercise/nutrition education, and behavioral health.
  Interventions: Behavioral: TLC Group Prenatal Care
- Traditional Prenatal Care (No Intervention): Subjects randomized to routine care will receive their prenatal care with their primary obstetric provider. Patients are seen for 10-15 minutes every four weeks until 28 weeks' gestation, every two weeks (or more by provider discretion) until 37 weeks and weekly until delivery. Visits focus on routine screening tests and prenatal care. Traditional care participants will receive a phone call once a month, until 28 weeks gestation, from a nurse practitioner to check-in on pregnancy goals, healthy eating, and exercise. Each subject's medical chart will be reviewed for demographics, antenatal management, maternal and neonatal outcomes.

INTERVENTIONS:
Behavioral: TLC Group Prenatal Care — TLC will start in the late first trimester or early second trimester and run for ~6-10 sessions. Groups of 2-10 consented women, with two or more GDM risk factors, will meet under the supervision of an obstetric provider (nurse practitioner or MD) and co-facilitator (health educator, nutritionist, or nurse) for two-hour sessions. A major focus of TLC will be education, and much of each visit will be spent on pregnancy, exercise/nutrition education, and behavioral health.
  Arms: TLC Group Prenatal Care

SUMMARY:
To conduct a randomized trial to determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal and neonatal outcomes in women at high risk for developing gestational diabetes mellitus (GDM).

DETAILED DESCRIPTION:
Long term, the investigator aims to test the central hypothesis that those in TLC will have better maternal and neonatal outcomes than those in TC. The objective is to conduct a randomized trial to determine the effect of TLC group prenatal care on birthweight and neonatal body composition, maternal healthy lifestyle and diabetes-related outcomes, delivery and neonatal outcomes, and psychosocial stress and depression.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* ≤16 weeks gestation
* Two or more of the following GDM risk factors:
* BMI ≥ 25
* Physical inactivity
* First degree relative with diabetes
* High risk race or ethnicity (African American, Latino, Native American, Asian American, Pacific Islander)
* Prior infant weighing ≥ 4,000 g
* Prior GDM
* Hypertension (140/90 mm Hg or receiving treatment)
* High-density lipoprotein cholesterol level <35 mg/dL or triglycerides > 250 mg/dL
* Polycystic ovarian syndrome
* A1c ≥ 5.7%
* Impaired glucose tolerance
* Impaired fasting glucose on previous testing
* History of cardiovascular disease
* Ability to attend group prenatal visits at specified days and times
* Willingness to be randomized
* Ability to give informed consent

Exclusion Criteria:

* Type 2 diabetes (eligible for Diabetes Group Care)
* Positive glucose challenge test during early pregnancy
* Multiple gestation (require extra care)
* Major fetal anomaly (require extra care)
* Serious medical co-morbidity necessitating more care than can be safely provided in group setting, as deemed by medical provider (require extra care)
* Serious psychiatric illness, including schizophrenia, necessitating more care than can be safely provided in group setting, as deemed by medical provider (require extra care)

Min Age: 13 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2019-11-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Effects of TLC group prenatal care on birth weight | Delivery/within 1 week of delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant weight in grams
Effects of TLC group prenatal care on neonatal length | Delivery/within 1 week of delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant length in cm
Effects on TLC group prenatal care on neonatal head circumference | Delivery/within 1 week of delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant head circumference in cm
Effects of TLC group prenatal care on infant skinfold thickness | Delivery/within 1 week of delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant skinfold thickness of ilium, thigh, triceps, and subscapular

SECONDARY OUTCOMES:
Maternal diagnosis of gestational diabetes | Up to the time of delivery
  Assessing maternal diagnosis of gestational diabetes using 2-step method(1-hour glucose challenge test, 3-hour glucose tolerance test, need for medication)
Physical activity and eating behavior | At enrollment, the last study visit/delivery, and 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on physical activity and eating behavior survey
Maternal gestational weight gain | Initial visit through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal gestational weight gain
Maternal hypertensive disorders of pregnancy including gestational hypertension, chronic hypertension, preeclampsia, eclampsia, and HELLP | Initial visit through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal hypertensive disorders of pregnancy
Rates of appointment attendance | Up to the time of delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on number of prenatal visits attended
Rates of maternal postpartum visit attendance for those in TLC compared to traditional prenatal care | 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on postpartum visit attendance
Rate of maternal contraception initiation for those in TLC compared to traditional prenatal care. | Delivery through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal postpartum contraception initiation
Breastfeeding rates among those in TLC compared to traditional prenatal care. | Delivery through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal breastfeeding
Postpartum weight retention | Up to 12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal postpartum weight retention
Postpartum 2 hour glucose tolerance testing (if applicable) | 4-12 weeks Postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal glucose tolerance testing
Insulin resistance | Through study completion, up to 12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal insulin resistance (fasting and 30 min insulin).
Insulin sensitivity | Through study completion, up to 12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal insulin sensitivity (fasting and 30 min insulin).
Assessing prenatal care patient satisfaction for those in TLC compared to traditional prenatal care using a satisfaction survey. | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal prenatal care satisfaction
Neonatal gestational age at delivery | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant gestational age at delivery
Induction of labor rates for those in TLC compared to traditional prenatal care | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal induction of labor
Mode of delivery for those in TLC compared to traditional prenatal care. | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC)on maternal mode of delivery
Neonatal shoulder dystocia rates for those in TLC compared to traditional prenatal care. | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant shoulder dystocia
Neonatal APGAR score | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant APGAR score
Neonatal cord blood analytes | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant cord blood analytes, c-peptide.
Neonatal cord blood analytes of pH for those in TLC compared to traditional prenatal care. | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant cord blood analytes, pH.
Neonatal cord blood analytes of base excess for those in TLC compared to traditional prenatal care. | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant cord blood analytes, base excess.
Neonatal NICU admission | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant NICU admission
Neonatal hypoglycemia | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant hypoglycemia
Neonatal hematocrit | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant hematocrit
Neonatal jaundice | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant jaundice
Neonatal respiratory distress syndrome | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant respiratory distress syndrome
Neonatal stillbirth | Delivery
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on infant stillbirth
Depression | Enrollment through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal depression using Edinburgh Postnatal Depression Scale
Psychosocial stress | Enrollment through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal stress using the perceived stress scale
Determine the effect of TLC on psychosocial stress and depression using the pregnancy distress questionnaire | Enrollment through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal distress
Determine the effect of TLC on psychosocial stress and depression using the life events checklist | Enrollment through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal life events
Determine the effect of TLC on psychosocial stress and depression using the generalized anxiety disorder-7 test | Enrollment through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal anxiety
Determine the effect of TLC on psychosocial stress and depression using the Munich Chronotype Questionnaire (MCTQ) | Enrollment through 4-12 weeks postpartum
  Determine the effect of Targeted Lifestyle Change Group Prenatal Care (TLC) on maternal sleep hygiene.

CONTACTS AND LOCATIONS:
Overall Officials: Ebony B Carter, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - Washington University in St. Louis, St Louis, Missouri
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina